CLINICAL TRIAL: NCT05651451
Title: Effect of Laser Acupuncture on Metabolic Syndrome in Obese Postmenopausal Women. A Randomized Controlled Study
Brief Title: Effect of Laser Acupuncture on Metabolic Syndrome in Obese Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 67
Record Dates: First submitted 2022-12-06; First posted 2022-12-15 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture group (Active Comparator): All women in group (B) were received 24 activated laser acupuncture treatments. Treatments was performed 3 times per week for 8 weeks.Laser acupuncture was applied withwavelength of 810 nm, power output of 150 mW in continuous wave mode and energy density laser of 4 J/cm2 with irradiation time 3 min/point. Total duration of the training session was 30 minutes.Before starting the first treatment session, each woman was instructed briefly about the nature of the treatment to gain her confidence and cooperation. The surface of the treated skin was cleaned with alcohol wipe in order to remove any material that could absorb or disperse the radiationon the surface.The laser handheld device (laser beam spot size ≤ 36 mm2) was applied directly and perpendicularly to avoid scattering the beam, The Laser probe was applied to the surface of skin before switching on apparatus.
  Interventions: Device: Laser acupuncture; Dietary Supplement: energy-restricted diet
- Diet regimen group (Active Comparator): All post-menopausal women followed an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E
  Interventions: Dietary Supplement: energy-restricted diet

INTERVENTIONS:
Device: Laser acupuncture — 24 activated laser acupuncture treatments. Treatments was performed 3 times per week for 8 weeks.Laser acupuncture was applied withwavelength of 810 nm, power output of 150 mW in continuous wave mode and energy density laser of 4 J/cm2 with irradiation time 3 min/point
  Arms: Laser acupuncture group
Dietary Supplement: energy-restricted diet — All post-menopausal women followed an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E

SUMMARY:
Thirty postmenopausal women were collected from outpatient clinic of faculty of physical therapy in Benha University to participate in this study. Their ages were ranged from 55-65 years old and their body mass index (BMI) ranged from 30 to 34.9 Kg/m2. They were divided randomly into 2 equal groups; Group A: received diet regimen, Group B: received diet regimen and treated with laser acupuncture for 30 minutes, 3 sessions per week for two months

DETAILED DESCRIPTION:
-Group A (control group): All post-menopausal women followed an energy-restricted diet for 8 weeks. Meal plan that creates an energy deficit of 500 to 1000 Kcal per day less than the individual's average daily intake was suitable for weight reduction.Each post-menopausal woman followed Dietary Approaches to Stop Hypertension (DASH) which : low in total fat, cholesterol, red meat, sweets and sugar containing beverages, emphasize fish, nuts, fruits, vegetables and whole grains and it also rich in Potassium(6900mg), Calcium(1200-1500mg) and Magnesium, as well as vitamins A, C and E.

II-Group B (study group):

All women in group (B) were received 24 activated laser acupuncture treatments. Treatments was performed 3 times per week for 8 weeks.Laser acupuncture was applied withwavelength of 810 nm, power output of 150 mW in continuous wave mode and energy density laser of 4 J/cm2 with irradiation time 3 min/point. Total duration of the training session was 30 minutes.Before starting the first treatment session, each woman was instructed briefly about the nature of the treatment to gain her confidence and cooperation. The surface of the treated skin was cleaned with alcohol wipe in order to remove any material that could absorb or disperse the radiationon the surface.The laser handheld device (laser beam spot size ≤ 36 mm2) was applied directly and perpendicularly to avoid scattering the beam, The Laser probe was applied to the surface of skin before switching on apparatus.

Laser acupuncture was applied on:

* Cv4 (Guanyuan) (3 cun inferior to the center of the umbilicus);
* Cv9 (Shuifen) (1 cun above the center of the umbilicus);
* Cv12 (Zhongwan) (4 cun above the center of the umbilicus);
* St25 (Tianshu) (2 cun lateral to the midline of the umbilicus);
* St36 (Zusanli) (one finger width lateral from the anterior crest of the tibia);
* Sp6 (Sanyinjiao) (3 cun directly above the tip of the medial malleolus);
* St40 (Fenglung) (8 cun superior to the tip of the external malleolus);
* LI4 (Hegu) (on the highest spot of the muscle when the thumb and index fingers are brought close together);
* LI11 (Quchi) (on the outside end of the crease on the elbow);
* and PC6 (Neiguan)( three finger breadths below the wrist on the inner forearm in between the two tendons.

ELIGIBILITY:
Inclusion Criteria:

* prehypertension and hypertension stage I
* overweight or obesity class I
* age 55 to 65 years

Exclusion Criteria:

* systolic blood pressure exceeding 159 mm Hg
* diastolic blood pressure exceeding 99 mm Hg,
* diabetic neuropathy disease,
* patients with mental or psychological disorders,
* skin disorders
* bleeding disorders
* musculoskeletal disorders

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Lipid profile TG | 8 weeks after treatment
  Triglycerides in mmol/L will be measured
Lipid profile HDL | 8 weeks after treatment
  High density lipoprotein in mmol/L will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No